CLINICAL TRIAL: NCT00607516
Title: Radiostereometric Analysis of Acetabular Wear and Periprosthetic Bone Mineral Density Changes in Cemented and Uncemented Hemiarthroplasties for Femoral Neck Fractures
Brief Title: Radiostereometric Analysis of Acetabular Wear and Periprosthetic Bone Mineral Density Changes in Hemiarthroplasties
Acronym: HEMI-RSADEXA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Lars Nordsletten, Ulleval university hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HEMI-RSA-DEXA; REK I (Norway) 151-05-04061
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2009-06-24 (Estimated); Status verified 2007-02

CONDITIONS: Femoral Neck Fractures; Bone Density; Acetabular Wear; Hemiarthroplasty
Keywords: fracture; arthroplasty; wear; osteoporosis; bone
MeSH Terms: conditions — Femoral Neck Fractures; Fractures, Bone; Osteoporosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cemented (Active Comparator): Cemented primary bipolar hemiarthroplasty of the hip
  Interventions: Procedure: Cemented primary bipolar hemiarthroplasty of the hip
- Uncemented (Active Comparator): Uncemented primary bipolar hemiarthroplasty of the hip
  Interventions: Procedure: Uncemented primary bipolar hemiarthroplasty of the hip

INTERVENTIONS:
Procedure: Cemented primary bipolar hemiarthroplasty of the hip — Cemented primary bipolar hemiarthroplasty of the hip
  Other Names: Spectron, Smith & Nephew, Memphis, TN
  Arms: Cemented
Procedure: Uncemented primary bipolar hemiarthroplasty of the hip — Uncemented primary bipolar hemiarthroplasty of the hip
  Other Names: Corail, DePuy/Johnson and Johnson, United Kingdom
  Arms: Uncemented

SUMMARY:
Substudy and continuation of HEMI-SAB-UUS (NCT00491673)

Study on radiostereometric measurements of acetabular wear in bipolar hemiarthroplasties and measurements of periprosthetic bone mineral density in cemented and uncemented hemiarthroplasties in patients with femoral neck fractures.

Null hypothesis: No difference in acetabular wear or in bone mineral density changes between cemented and uncemented hemiarthroplasties

DETAILED DESCRIPTION:
Patients are randomised to treatment with cemented or uncemented bipolar hemiarthroplasty. 1mm tantalum markers are inserted in the pelvis during surgery. RSA X-rays and DEXA measurements conducted postoperatively, after 3 and 12 months. Follow-up visits and clinical examination at 3 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Femoral neck fracture
* 65 years or older
* Able to walk independently

Exclusion Criteria:

* Cognitive dysfunction
* Infection
* Fracture caused by malignant disease

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-03; Primary Completion 2009-01 (Estimated); Study Completion 2009-01 (Estimated)

PRIMARY OUTCOMES:
Acetabular wear in mm | 1 year
Loss of bone mineral density (BMD) | 1 year

SECONDARY OUTCOMES:
Functional outcome including pain (Harris Hip Score) | 1 year
Activities Of Daily Living (Barthels ADL-Index) | 1 year
Quality Of Life (EQ-5D) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lars Nordsletten, Prof MD PhD, Study Director — Ullevål University Hospital, University of Oslo
Locations (1):
- Ullevål University Hospital, Oslo, Oslo County, Norway